CLINICAL TRIAL: NCT03651934
Title: Verification of Correlation Between Genetic Testing of Nutritional Metabolism and Clinical Biochemical Indicators
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Liuyanping, Clinical Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hs-1646
Record Dates: First submitted 2018-08-06; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Pregnant Women

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal iron (Experimental)
  Interventions: Dietary Supplement: Normal iron; Dietary Supplement: Weak iron
- Weak iron (Experimental)
  Interventions: Dietary Supplement: Normal iron; Dietary Supplement: Weak iron
- Normal selenium (Experimental)
  Interventions: Dietary Supplement: Normal selenium; Dietary Supplement: Weak selenium
- Weak selenium (Experimental)
  Interventions: Dietary Supplement: Normal selenium; Dietary Supplement: Weak selenium

INTERVENTIONS:
Dietary Supplement: Normal iron — The intervention was divided into two stages, the first stage lasted for 4 weeks, and the dosage used was the dietary nutrient recommendation amount, namely the dietary recommendation amount standard for early pregnancy (iron 20mg/d), and the middle stage of pregnancy (iron 24mg/d). The second stage lasts for 4 weeks. For subjects in iron deficiency, the maximum tolerable amount (iron 42mg/d) is used for intervention. For those with good nutritional status, the dietary recommendation amount is maintained.
  Arms: Normal iron; Weak iron
Dietary Supplement: Weak iron — The intervention was divided into two stages, the first stage lasted for 4 weeks, and the dosage used was the dietary nutrient recommendation amount, namely the dietary recommendation amount standard for early pregnancy (iron 20mg/d), and the middle stage of pregnancy (iron 24mg/d). The second stage lasts for 4 weeks. For subjects in iron deficiency, the maximum tolerable amount (iron 42mg/d) is used for intervention. For those with good nutritional status, the dietary recommendation amount is maintained.
  Arms: Normal iron; Weak iron
Dietary Supplement: Normal selenium — The intervention was divided into two stages, the first stage lasted for 4 weeks, and the dosage used was the dietary nutrient recommendation amount, namely the dietary recommendation amount standard for early pregnancy (selenium 60ug/d), and the middle stage of pregnancy (selenium 65ug/d). The second stage lasts for 4 weeks. For subjects in selenium deficiency, the maximum tolerable amount (selenium 400ug/d) is used for intervention. For those with good nutritional status, the dietary recommendation amount is maintained.
  Arms: Normal selenium; Weak selenium
Dietary Supplement: Weak selenium — The intervention was divided into two stages, the first stage lasted for 4 weeks, and the dosage used was the dietary nutrient recommendation amount, namely the dietary recommendation amount standard for early pregnancy (selenium 60ug/d), and the middle stage of pregnancy (selenium 65ug/d). The second stage lasts for 4 weeks. For subjects in selenium deficiency, the maximum tolerable amount (selenium 400ug/d) is used for intervention. For those with good nutritional status, the dietary recommendation amount is maintained.
  Arms: Normal selenium; Weak selenium

SUMMARY:
The research plan is divided into two parts. The first part is the correlation study .It is planned to include women who prepare for pregnancy or in the early stages of pregnancy to carry out the detection of 25 loci SNP of 21 genes of 9 nutrients, to predict the nutritional abnormalities of 9 nutrients, and to determine the nutritional status of 9 nutrients, and then verify the correlation between nutrient metabolism related gene SNP and nutrient nutrition status .The second part selects iron and selenium which are commonly lacking in Chinese women of childbearing age. A intervention study is designed for these two nutrients. According to the SNP grouping of related gene loci, observe the effect of nutrition intervention and explore the nutrition intervention strategies of different SNP individuals.

ELIGIBILITY:
Inclusion Criteria:

* preparing for pregnancy or early pregnancy women (< 12w)
* no major surgery, trauma, or important viscera disease
* no long-term medication history
* No serious mental and psychological behavior abnormalities
* resident in Beijing, can accept regular prenatal in Beijing area
* signed informed consent

Exclusion Criteria:

* have taken medications that may affect the metabolism of nutrients, but are unable to provide their ingredients or doses, making it difficult to judge their effects
* From the first three months of this pregnancy to the time of inclusion, taking drugs that interfere with the absorption, metabolism, and utilization of nutrients.
* From the first three months of this pregnancy to the time of inclusion, Pregnant woman took iron, selenium, vitamin B6, vitamin B12, vitamin D preparations, and the dosage was higher than the corresponding physiological standard.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-10 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between the results of nutritional evaluation of selenium-related genes and selenium levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of selenium gene monitoring and the levels of selenium in vivo
Correlation between the results of nutritional evaluation of iron-related genes and iron levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of iron gene monitoring and the levels of iron in vivo
Correlation between the results of nutritional evaluation of vitamin B6-related genes and vitamin B6 levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of vitamin B6 gene monitoring and the levels of vitamin B6 in vivo
Correlation between the results of nutritional evaluation of vitamin B12-related genes and vitamin B12 levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of vitamin B12 gene monitoring and the levels of vitamin B12 in vivo
Correlation between the results of nutritional evaluation of vitamin D-related genes and vitamin D levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of vitamin D gene monitoring and the levels of vitamin D in vivo
Correlation between the results of nutritional evaluation of pantothenic acid-related genes and pantothenic acid levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of pantothenic acid gene monitoring and the levels of pantothenic acid in vivo
Correlation between gestational diabetes-related gene monitoring results and glycosylated hemoglobin，fasting blood glucose, fasting insulin levels in vivo | lasted for 4 weeks
  The correlation between the nutrition evaluation results of gestational diabetes-related gene monitoring and the levels of glycosylated hemoglobin，fasting blood glucose, fasting insulin in vivo
Correlation between gestational hypertension-related gene monitoring results and homocysteine, serum folic acid and RBC Folate levels in vivo | lasted for 4 weeks
  TThe correlation between the nutrition evaluation results of gestational hypertension-related gene monitoring and the levels of homocysteine, serum folic acid and RBC Folate in vivo
Correlation between hyperlipidemia-related gene monitoring results and the level of plasma lipid in vivo. | lasted for 4 weeks
  The correlation between the nutrition evaluation results of hyperlipidemia-related gene monitoring and the levels of plasma lipid in vivo
nutritional status | lasted for 4 weeks
  The nutritional status of selenium was compared between the normal selenium and week selenium group; The nutritional status of iron was compared between the normal iron and the weak group. Meanwhile, compare the selenium and iron nutritional status of the four groups before and after the intervention.

REFERENCES:
- [Derived] Zhao R, An Z, Sun Y, Xia L, Qiu L, Yao A, Liu Y, Liu L. Metabolic profiling in early pregnancy and associated factors of folate supplementation: A cross-sectional study. Clin Nutr. 2021 Sep;40(9):5053-5061. doi: 10.1016/j.clnu.2021.01.012. Epub 2021 Jan 23. PMID 34455263